CLINICAL TRIAL: NCT01096797
Title: Prospective Cohort Study Evaluating Incidence and Correlation Between Pain and Emergence Delirium After Adenotonsillectomy in Preschool Children
Brief Title: Correlation Between Pain and Emergence Delirium After Adenotonsillectomy in Preschool Children
Acronym: e-PONB ENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: San Gerardo Hospital (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Pablo Mauricio Ingelmo, U.O. Anestesia e Rianimazione I. San Gerardo Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AR-HSG 02-2009
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2009-11

CONDITIONS: Adenotonsillectomy; Postoperative Pain; Emergence Delirium
MeSH Terms: conditions — Pain, Postoperative; Emergence Delirium | interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children undergoing adenotonsillectomy (Experimental): Children between 2-6 years old undergoing elective adenoidectomy with or without tonsillectomy from the ENT Service of the San Gerardo Hospital.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — * Anaesthesia induction: sevoflurane 4 to 6% by mask and IV propofol 2-6 mg/kg.
  * Anaesthesia maintenance: sevoflurane 2-3 %
  * Intraoperative and postoperative analgesia: IV fentanyl 1,5-2,5 mcg/kg, IV paracetamol 15 mg/kg
  * Prevention of postoperative nausea and vomiting: dexamethasone 0,1 mg/kg, ondansetron 0,1 mg/kg

SUMMARY:
The purpose of this study is to determine the incidence of pain, emergence delirium and the combination of those postoperative negative behaviours during the first 15 minutes after awakening from sevoflurane anesthesia in pre-school children. Additionally this study will evaluate the relationship between emergence delirium and postoperative pain behaviour after adenotonsil surgery.

DETAILED DESCRIPTION:
Tonsillectomy and/or adenoidectomy is the most common surgery performed in paediatric population. Sevoflurane is the most frequently volatile anaesthetic used in paediatric population. It is well tolerated, allows rapid anaesthesia induction, faster emergence, orientation. A child who emerges from sevoflurane anaesthesia may experience a variety of behavioural disturbances described as "emergence delirium" (ED).

ED has been described as "a mental disturbance during the recovery from general anaesthesia consisting of hallucinations, delusions and confusion manifested by moaning, restlessness, involuntary physical activity, and thrashing about in bed" in the immediate post anaesthesia period. Additionally paranoid ideation has been observed in combination with these emergence behaviours.

Restless recovery from anaesthesia is an important problem. It may lead, along with injury to the child, bleeding from surgical site, to accidental removal of IV catheters and drains. Once ED occur, extra nursing care may be necessary, as well as supplemental sedative and/or analgesic medications, which may be associated to respiratory depression or airway obstruction and may delay patient discharge. Although long-term psychological implications of ED remain unknown, children with restless recovery from anaesthesia are seven times more likely to have new-onset separation anxiety, apathy, eating and sleep problems.

ED after sevoflurane anaesthesia has been suggested both to be and not to be associated with postoperative pain behaviour. Accordingly, adequate pain relief has been found to reduce or have no effect on ED after sevoflurane anaesthesia. Because a self-evaluation is difficult In preschool boy observational scales based on behaviour like CHIPPS, FLACC or CHEOPS are used for the measurement of pain.

Given that the child's behaviour evaluation at emergence is made with observational scales, a superimposition between ED and pain measurement is possible. Nurses and doctors using behavioural scales for the evaluation of ED and pain may not be able to differentiate pain from ED during awakening. This may led to the treatment of an autolimitated disturb (ED) or to the under treatment of pain after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female children from 2 to 6 years of age
* American Society of Anaesthesiologists Classification (ASA) I: without systemic disease
* American Society of Anaesthesiologists Classification (ASA) II: moderate systemic disease
* Scheduled for elective tonsillectomy and/or adenoidectomy.
* Children whose parents (or legal tutors) have given their informed written consent

Exclusion Criteria:

* Emergency surgery.
* Children whose parents (or legal tutors) denied their own consensus
* Children with known cognitive impairment
* A story of kidney, liver, pulmonary or cardiac disease.
* A history of chronic pain or use of analgesic drugs.
* Familiar or personal history of malignant hyperthermia
* Need premedication or total intravenous anaesthesia.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Emergence delirium evaluation: Pediatric Anesthesia Emergence Delirium scale (PAED) | First 15 minutes after awakening.
  Pediatric Anesthesia Emergence Delirium scale(PAED):The PAED scale consists of five psychometric items. To each of them it's possible to assign a score from 0 to 4 (maximum score 20 points). Emergence delirium was defined as a PAED scale score of 10 points of grater.
Pain: Face, Legs, Activity, Cry, Consolability Scale (FLACCS); Children and Infants Postoperative Pain Scale (CHIPPS); Children Hospital of Eastern Ontario Pain Scale (CHEOPS) | 15 minutes after awakening
  * FLACCS: five behavioural items scale with a maximum score of 10 points. Significant pain behaviour correspond to a FLACCS score of 4 points or greater.
  * CHIPPS: five behavioural items scale with a maximum score of 10 points. Significant pain behaviour correspond to a FLACCS score of 4 points or greater.
  CHEOPS: five behavioural items scale with a maximum score of 13 points. Significant pain behaviour correspond to a CHEOPS score of 7 points or greater

SECONDARY OUTCOMES:
Age
  Age groups: 2 to 4 ys and 5 to 6 ys
Time of exposure to sevoflurane
Awakening time
  Time between end of sevoflurane exposure and extubation

CONTACTS AND LOCATIONS:
Overall Officials: Pablo M Ingelmo, MD, Principal Investigator — Department of anesthesiology and resuscitation I, San Gerardo Hospital
Locations (1):
- Department of Perioperative Medicine and Intensive Care. San Gerardo Hospital, Monza, MB, Italy

REFERENCES:
- [Background] Holzki J, Kretz FJ. Changing aspects of sevoflurane in paediatric anaesthesia: 1975-99. Paediatr Anaesth. 1999;9(4):283-6. doi: 10.1046/j.1460-9592.1999.00415.x. No abstract available. PMID 10411761
- [Result] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Result] Vlajkovic GP, Sindjelic RP. Emergence delirium in children: many questions, few answers. Anesth Analg. 2007 Jan;104(1):84-91. doi: 10.1213/01.ane.0000250914.91881.a8. PMID 17179249
- [Result] Voepel-Lewis T, Malviya S, Tait AR. A prospective cohort study of emergence agitation in the pediatric postanesthesia care unit. Anesth Analg. 2003 Jun;96(6):1625-1630. doi: 10.1213/01.ANE.0000062522.21048.61. PMID 12760985
- [Result] Dahmani S, Stany I, Brasher C, Lejeune C, Bruneau B, Wood C, Nivoche Y, Constant I, Murat I. Pharmacological prevention of sevoflurane- and desflurane-related emergence agitation in children: a meta-analysis of published studies. Br J Anaesth. 2010 Feb;104(2):216-23. doi: 10.1093/bja/aep376. Epub 2010 Jan 3. PMID 20047899